CLINICAL TRIAL: NCT04720287
Title: Ultrasound Guided Quadratus Lumborum Block Compared to Caudal Bupivacaine/ Neostigmine in Pediatric Lower Abdominal Surgeries, a Randomized Controlled Trial
Brief Title: Ultrasound Guided Quadratus Lumborum Block Compared to Caudal Bupivacaine/ Neostigmine in Pediatric Lower Abdominal Surgeries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dr.Ibrahim Mamdouh Esmat, Assistant Professor of Anesthesia and Intensive Care Department, Faculty of Medicine, Ain- shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU MS 728/2020/2021
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Postoperative Analgesia
MeSH Terms: interventions — Bupivacaine; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1(QL group) (Active Comparator)
  Interventions: Drug: bupivacaine/ neostigmine.
- Group 2 (CB group) (Active Comparator)
  Interventions: Drug: bupivacaine/ neostigmine.

INTERVENTIONS:
Drug: bupivacaine/ neostigmine. — will receive bilateral ultrasound guided QLB
  Arms: Group 1(QL group)
Drug: bupivacaine/ neostigmine. — will receive ultrasound guided CB.
  Arms: Group 2 (CB group)

SUMMARY:
The aim of this study is to compare the postoperative pain control in children undergoing lower abdominal surgeries receiving QL block with those receiving caudal bupivacaine/ neostigmine.

ELIGIBILITY:
Inclusion Criteria:

* Patients American Society of Anesthesiologists physical status (ASA) I or II.
* Consent from parents or legal guardian(s).
* Lower abdominal surgeries.

Exclusion Criteria:

* Parents' refusal or legal guardian's refusal.

  * Infection at the injection site.
  * Known allergy to bupivacaine and/or neostigmine.
  * Contraindications to regional anesthesia (including coagulopathy and local infection).
  * Anatomical anomalies at the site of the block.

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
The total amount of paracetamol doses (mg) | 24 hours postoperatively
  The total amount of paracetamol doses (mg)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No